CLINICAL TRIAL: NCT05058768
Title: Exosomes in Urine, Blood, and Alveolar Lavage Fluid From Patients With Acute Respiratory Distress Syndrome (ADRS) Were Sequenced by Omics
Brief Title: Omics Sequencing of Exosomes in Body Fluids of Patients With Acute Lung Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-143
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2021-09

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine or alveolar lavage fluid samples of the experimental group and the control group were reserved for omics sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Healthy people served as the control group
- experimental group: Patients with acute lung injury were treated as the experimental group.
  Interventions: Diagnostic Test: The lungs causes and extrapulmonary factors

INTERVENTIONS:
Diagnostic Test: The lungs causes and extrapulmonary factors — Acute lung injury due to internal and external pulmonary causes can be used as intervention items in this study, and intervention items can be excluded according to inclusion criteria and exclusion criteria.
  Groups: experimental group

SUMMARY:
The exosomes in the experimental group and the control group were sequenced to find the difference of the two groups, providing a basis for subsequent basic research.

DETAILED DESCRIPTION:
This study is an observational study, mainly collected by infection, trauma, burns and other non cardiac causes without any related comprehensive character drug treatment of acute respiratory distress (ARDS) in patients with blood, urine or alveolar lavage fluid specimens, used to extract exosomes for omics sequencing, relevant histomorphic variations in exosomes of this disease were obtained, In addition, functional verification of genes or proteins with different changes will be carried out to provide clinical basis for subsequent basic research.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of experimental group:

* Signed informed consent voluntarily;
* Age: >18 years old, gender: no restrictions ;
* Patients with known clinical manifestations of respiratory impairment or new/aggravated respiratory symptoms diagnosed within one week of onset according to the Berlin definition guidelines.

Control group inclusion criteria:

* Age ≥18 years old (including 18 years old), male and female;
* Male weight ≥50 kg, female weight ≥45kg, and body mass index (BMI) between 19 and 26(inclusive), BMI= weight (kg)/ height (㎡);
* No smoking, alcohol addiction, no history of drug abuse;
* No diabetes, asthma, copd, chronic renal insufficiency and other basic diseases; No history of major diseases or infectious diseases (including hepatitis B, hepatitis C, HIV, syphilis);
* Those who have not taken drugs recently.

Exclusion Criteria:

Exclusion criteria of experimental group:

* Patients with diabetes, chronic renal insufficiency, malignant tumors and other basic diseases;
* severe malnutrition;
* Pregnant or lactating women;
* The researcher judged that he was not suitable to participate in this study.

Exclusion criteria for the control group:

* pregnant or lactation women;
* severe malnutrition;
* The researcher judged that he was not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The experimental group was patients with acute lung injury, which was caused by various direct and indirect injury factors of alveolar epithelial cells and capillary endothelial cells, resulting in diffuse pulmonary interstitial and alveolar edema, resulting in acute hypoxic respiratory insufficiency. The control group was healthy subjects.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-05-06 (Estimated); Primary Completion 2023-05-07 (Estimated); Study Completion 2024-12-16 (Estimated)

PRIMARY OUTCOMES:
Compare the omics differences of blood samples between the experimental and control groups | one year
  Collected separately in the experimental group and the control group participants' blood as a specimen, It is used to obtain exosomes and perform omics sequencing, to obtain the histopathological differences of exosomes between experimental and control groups, In addition, functional verification of genes or proteins with different changes will be carried out to provide clinical basis for subsequent basic research .
Compare the omics differences of urine samples between the experimental and control groups | one year
  Collected separately in the experimental group and the control group participants' urine as a specimen, It is used to obtain exosomes and perform omics sequencing, to obtain the histopathological differences of exosomes between experimental and control groups, In addition, functional verification of genes or proteins with different changes will be carried out to provide clinical basis for subsequent basic research .

SECONDARY OUTCOMES:
Compare the omics differences of alveolar lavage fluid samples between the experimental and control groups | one year
  Collected separately in the experimental group and the control group participants' alveolar lavage fluid as a specimen, It is used to obtain exosomes and perform omics sequencing, to obtain the histopathological differences of exosomes between experimental and control groups, In addition, functional verification of genes or proteins with different changes will be carried out to provide clinical basis for subsequent basic research .

CONTACTS AND LOCATIONS:
Overall Officials: linzhong yu, professor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No